CLINICAL TRIAL: NCT00005480
Title: Cardiovascular Disease Knowledge/Morbidity--Socioeconomic Cohort Outcomes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4964; R03HL057578 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To elucidate the interrelationship of level of cardiovascular disease knowledge and subsequent clinical health status by merging population-based cardiovascular disease risk factor survey data with patient-level hospital data. The overall goal was to assess outcomes in the positive/negative association between level of cardiovascular disease knowledge and incidence and relative degree of morbidity among a cohort with and without major cardiovascular disease risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Evidence shows a growing disparity in the prevalence of modifiable risk factors and incidence of cardiovascular disease between upper and lower socioeconomic status (SES) individuals. Trends in knowledge about risk factors and risk reduction strategies parallel these findings. Research determining the differential association between level of cardiovascular disease knowledge and subsequent clinical health status had not been conducted.

DESIGN NARRATIVE:

Analyses were stratified according to SES (via years of formal education), controlling for age, gender, and ethnicity (Latino/Anglo). Sociodemographic, physiologic, and knowledge measurements were available on each participant. Morbidity estimates and clinical health status indicators were available via primary and secondary discharge diagnostic codes from public-use hospital discharge databases collected on all California hospital admissions for the entire study period. The Stanford Five City Program data were merged with the hospital discharge data, matching on survey participant's social security number which was subsequently converted to a unique personal identifier. Baseline 1989/90 and 1991 through 1995 longitudinal outcomes were assessed.

There were three main aims, all of which had epidemiologic and cardiovascular disease health policy prevention implications: Aim 1: Characterize the distribution of hospitalized versus non-hospitalized SES sub-cohorts according to level of C.D. knowledge, physiologic risk factor prevalence, and clinical morbidity prevalence. Aim 2: Test the hypothesis that morbidity differences between hospitalized SES sub-cohorts would vary as a function of baseline level of cardiovascular disease knowledge and risk factor prevalence. Aim 3: Test the hypothesis that morbidity would rise among hospitalized lower SES sub-cohorts, resulting in widening health status disparities by the end of the study period. Parametric and nonparametric analytic methods were used, including analysis of variance and covariance, and various regression techniques.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 1998-08 (Actual)